CLINICAL TRIAL: NCT03694964
Title: Effects of Oral Citrulline Supplementation in Sarcopenia for Patients With Severe Chronic Respiratory Failure by COPD
Brief Title: Severe Chronic Respiratory Failure and Citrulline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 38RC17.310
Record Dates: First submitted 2018-06-06; First posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Sarcopenia; Citrulline; Body composition; Denutrition
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sarcopenia

STUDY DESIGN:
Intervention Model Description: After signing the informed consent form, the patients will be randomized either in the experimental group (Citrulline (ProteiCIT®): 10 g / day) or in the control group (placebo).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind study: treatment (experimental group) vs placebo (control group).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementation with Citrulline (Experimental): Patients will receive citrulline (ProteoCIT®) 10 mg by day during 45 days
  Interventions: Drug: ProteoCIT®
- Placebo (Placebo Comparator): Patients will receive placebo (one tablet by day) during 45 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: ProteoCIT® — 30 patients will be randomized into the group that will receive 10 mg of citrulline and 30 patients will be randomized into the placebo group for 45 days
  Arms: Supplementation with Citrulline
Drug: Placebo Oral Tablet — 30 patients will be randomized into the group that will receive 10 mg of citrulline and 30 patients will be randomized into the placebo group for 45 days
  Arms: Placebo

SUMMARY:
Because of its very high bioavailability and its specific and direct action on protein synthesis, the investigators hypothesize that citrulline supplementation would be an innovative nutritional strategy to improve the peripheral muscle mass and strength in COPD patients with severe chronic respiratory failure.

This supplementation would be more effective if the pathology is severe and the chronic systemic inflammation important. The benefits of this supplementation could help the most severe patients break out of the cycle of inactivity and thus optimize their quality of life.

The main objective of this study is to evaluate the impact of 45-day nutritional supplementation with Citrulline (10 g / day) on the body composition (lean body mass) in malnourished COPD patients with severe chronic respiratory failure.

DETAILED DESCRIPTION:
Denutrition in patients with COPD (Chronic Obstructive Pulmonary Disease) is characterized by muscle atrophy and loss of strength in the lower extremities. It worsens the symptomatology, exercise intolerance, impaired quality of life and prognosis of patients.

Consequence of a protein deficiency associated with systemic inflammation, denutrition is becoming increasingly important in patients with chronic respiratory failure (CRF). L-citrulline is an amino acid having a direct action on muscle protein synthesis. The citrulline supplementation is an effective treatment to fight against muscle loss in aging subjects. Its impact on the functional and nutritional status of COPD patients has not been studied.

Our main objective is to determine the impact of supplementation with Citrulline on mass and peripheral muscle strength in COPD with CRF. Our secondary objectives are to identify whether these benefits are dependent on the severity of the disease and if they are associated with increased physical activity, exercise tolerance and an improvement in symptoms and quality of life. This prospective, randomized, controlled, double-blind study will include 60 stable COPD patients (stage 3 and 4), with long-term oxygen therapy and / or non-invasive ventilation, BMI <25 kg.m2 and suspicion of sarcopenia.

For 45 days, patients will receive either citrulline (ProteoCIT®, 10mg) or placebo. The severity of COPD will be assessed by spirometry and blood gas data, the BODE index, exacerbations, comorbidities, nutritional status and systemic inflammation (CRPs, Fibrinogens). the investigators will evaluate before and after supplementation: body composition (DEXA), quadriceps strength and grip strength, walking speed, the exercise tolerance (6MWD), dyspnea (MMRC scales, BDI / TDI), quality of life (CAT and VSRQ questionnaires). Physical activity will be assessed by continuous actigraphy. This multicenter study will be conducted in 3 French hospitals: Grenoble, Nancy, Dijon.

ELIGIBILITY:
Inclusion Criteria:

* COPD Gold III and IV
* involuntary decrease in weight ≥ 5% in the last 6 months,
* BMI < 25 kg.m²
* suspicion of sarcopenia marked by a score higher than 4 on the SARC-F questionnaire
* clinical stability defined by no exacerbation requiring hospitalization for at least 3 months
* long-term oxygen therapy (≥ 12h / day) and / or non-invasive ventilation for at least 6 months
* At least one exacerbation requiring hospitalization in the year before inclusion.
* Informed consent written

Exclusion Criteria:

* Restrictive or mixed respiratory disease.
* Long-term systemic corticosteroids (> 6 months per year)
* Severe and terminal renal failure (creatinine clearance <30ml / min)
* Patients with severe hypotension, uncontrolled hypertension
* Contraindication to taking citrulline: anticoagulant and anticancer chemotherapy
* Osmotic diarrhea
* Taking food supplements whatever its form.
* Severe and / or unbalanced progressive disease that may be life-threatening in the medium term,
* Proven psychiatric pathology (schizophrenia type, dementia, bipolar / severe psychotic disorders, severe depressive syndrome),
* Cognitive or psychomotor problem that limit the realization and understanding of the different evaluations,
* Simultaneous participation in another research involving the human person
* Pregnant, parturient or breastfeeding women
* deprivation of liberty by judicial or administrative decision, protection by law, under the protection of justice, under guardianship or trusteeship,
* No affiliation to a social security scheme.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Impact of a 45-day nutritional supplementation with Citrulline (10 g / day) on body composition (lean body mass) of malnourished patients with COPD and severe chronic respiratory failure | 45 days
  Lean mass (kg.m-2) measured by DEXA

SECONDARY OUTCOMES:
Impact of a nutritional supplementation with Citrulline on body composition | 45 days
  Regional variations of fat and bone mass measured by DEXA
Impact of a nutritional supplementation with Citrulline on muscular force | 45 days
  Grip force, Maximum strength of the quadriceps
Impact of a nutritional supplementation with Citrulline on tolerance to effort | 45 days
  3 min chair test
Impact of a nutritional supplementation with Citrulline on BODE stage | 45 days
  BODE score - The BODE score is composed of the following parameters: the body mass index, the post-bronchodilator FEV1 expressed as a percentage of the theoretical values (airflow obstruction), the dyspnoea score measured by the modified scale of the RCM ( Dyspnea) and the distance in meters traveled during a 6-minute walk test (Exercise).Each value of each parmeter corresponds to 1 point (from 0 to 4) and we add everything. The results are: score 0 to 2: mortality 15% at 4 years; and score 7 to 10: 80% mortality at 4 years
Impact of a nutritional supplementation with Citrulline on inflammation and nutritional status | 45 days
  BMI
Impact of a nutritional supplementation with Citrulline on quality of life and dyspnea | 45 days
  Quality of life questionaries: COPD assessement Test (CAT): the participants answers differents questions that make it possible to measure the state of health of the patient.
Impact of a nutritional supplementation with Citrulline on physical activity | 45 days
  Actigraphy
Impact of a nutritional supplementation with Citrulline on tolerance to effort | 45 days
  Pulmonary function test
Impact of a nutritional supplementation with Citrulline on tolerance to effort | 45 days
  Exacerbation number
Impact of a nutritional supplementation with Citrulline on tolerance to effort | 45 days
  Comorbidities
Impact of a nutritional supplementation with Citrulline on tolerance to effort | 45 days
  Blood gas results
Impact of a nutritional supplementation with Citrulline on quality of life and dyspnea | 45 days
  Quality of life questionaries: Visual Simplified respiratory questionary (VSRQ)
Impact of a nutritional supplementation with Citrulline on quality of life and dyspnea | 45 days
  Quality of life questionaries: Medical Research Council (mMRC)
Impact of a nutritional supplementation with Citrulline on quality of life and dyspnea | 45 days
  Quality of life questionaries: The baseline and Transition Dyspnea Indices (TDI/BDI scale)
Impact of a nutritional supplementation with Citrulline on quality of life and dyspnea | 45 days
  Quality of life questionaries: Disability Related to COPD tool (DIRECT) : a self-administered questionnaire designed to evaluate the impact of COPD on the patient's daily activities
Impact of a nutritional supplementation with Citrulline on inflammation and nutritional status | 45 days
  MNA test : Mini Nutritional Assessment
Impact of a nutritional supplementation with Citrulline on inflammation and nutritional status | 45 days
  a blood sample will be taken from the participants to measure the effects of citrulline on the inflammation and nutritional status of the patient. C reactive protein (CRPus), inflammation marker
Impact of a nutritional supplementation with Citrulline on inflammation and nutritional status | 45 days
  Fibrinogen : inflammation marker that will be measured on a blood sample.
Impact of a nutritional supplementation with Citrulline on inflammation and nutritional status | 45 days
  Transthyretinemia biological parameter that will measure the nutritional status of the patient.will be mesasured on blood sample.
Impact of a nutritional supplementation with Citrulline on inflammation and nutritional status | 45 days
  Albuminemia : biological parameter that will measure the nutritional status of the patient.will be mesasured on blood sample.
Impact of a nutritional supplementation with Citrulline on inflammation and nutritional status | 45 days
  glycemia biological parameter that will measure the nutritional status of the patient.will be mesasured on blood sample.
Impact of a nutritional supplementation with Citrulline on inflammation and nutritional status | 45 days
  Insulinemia biological parameter that will measure the nutritional status of the patient. will be mesasured on blood sample.
Impact of a nutritional supplementation with Citrulline on inflammation and nutritional status | 45 days
  Acid-aminemia biological parameter that will measure the nutritional status of the patient. will be mesasured on blood sample.
Impact of a nutritional supplementation with Citrulline on inflammation and nutritional status | 45 days
  3 MethylHistine / urinary creatinine : this biological parameter will be measure on the urine: biological parameter measured on the urine. which will help to highlight the nutritional status of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: CHRISTOPHE PISON, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - Hôpital François Mitterrand - CHU de Dijon, Dijon
  - Hôpitaux de Brabois - CHU de Nancy, Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schols AM, Ferreira IM, Franssen FM, Gosker HR, Janssens W, Muscaritoli M, Pison C, Rutten-van Molken M, Slinde F, Steiner MC, Tkacova R, Singh SJ. Nutritional assessment and therapy in COPD: a European Respiratory Society statement. Eur Respir J. 2014 Dec;44(6):1504-20. doi: 10.1183/09031936.00070914. Epub 2014 Sep 18. PMID 25234804
- [Background] Cano NJ, Roth H, Court-Ortune I, Cynober L, Gerard-Boncompain M, Cuvelier A, Laaban JP, Melchior JC, Pichard C, Raphael JC, Pison CM; Clinical Research Group of the Societe Francophone de Nutrition Enterale et Parenterale. Nutritional depletion in patients on long-term oxygen therapy and/or home mechanical ventilation. Eur Respir J. 2002 Jul;20(1):30-7. doi: 10.1183/09031936.02.01812001. PMID 12166577
- [Background] Woo J, Leung J, Morley JE. Validating the SARC-F: a suitable community screening tool for sarcopenia? J Am Med Dir Assoc. 2014 Sep;15(9):630-4. doi: 10.1016/j.jamda.2014.04.021. Epub 2014 Jun 16. PMID 24947762